CLINICAL TRIAL: NCT05407571
Title: Clinical Significance of Echogenic Amniotic Fluid on Perinatal Outcome
Brief Title: Echogenic Amniotic Fluid on Perinatal Outcome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Egymedicalpedia (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Supportive Care
Other Study IDs: Hanaa Ibrahim
Record Dates: First submitted 2022-05-29; First posted 2022-06-07 (Actual); Last update posted 2023-09-08 (Actual); Status verified 2023-09

CONDITIONS: Amniotic Fluid; Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Echogenic Amniotic Fluid (Other): estimation the nature of echogenic amniotic fluid.to overcome unnecessary intervention due to turbid amniotic fluid, assessing the neonatal outcome and estimation the gestational age at time of delivery in patients with echogenic amniotic fluid.
  Interventions: Behavioral: Significance of Echogenic Amniotic Fluid on Perinatal Outcome

INTERVENTIONS:
Behavioral: Significance of Echogenic Amniotic Fluid on Perinatal Outcome — To estimate the nature of echogenic amniotic fluid.and To overcome unnecessary intervention due to turbid amniotic fluid, assess neonatal outcome and estimate gestational age at time of delivery in patients with echogenic amniotic fluid.

SUMMARY:
Amniotic fluid is the liquid that surrounds a developing fetus in the amniotic sac and is usually clear to pale yellow in color. Amniotic fluid composition is complex with many maternal and fetal constituents. It is mainly formed from fetal plasma volume, fetal urine, fetal respiratory system, gastrointestinal tract, umbilical cord, and fetal surface of the placenta. The composition of the Amniotic fluid changes with the gestational age with an average pH of 7.2 and specific gravity of 1.0069-1.008

DETAILED DESCRIPTION:
The sonographic appearance of amniotic fluid has been described as both anechoic and echogenic. The clinical significance of echogenic amniotic fluid remains undetermined. Increased echogenicity of the amniotic fluid may represent meconium. The presence of echogenic amniotic fluid at term on sonography is uncommon. The presence of meconium, blood or vernix caseosa in amniotic fluid may cause echogenicity.

The existence of meconium in amniotic fluid raises concerns about fetal well-being, the ability of the fetus to tolerate labor, or, most importantly, the risk of fetal/ neonatal demise . For these reasons, obstetricians tend to increase the frequency of prenatal visits to assess fetal well-being with non-stress tests or biophysical profiles (when there is no other indication for them), and even to induce labor when amniotic fluid is echogenic. On the other hand, elective induction of labor at term carries risks such as increased rate of cesarean section, uterine rupture or unexpected neonatal prematurity.

The presence of echogenic and dense particles in amniotic fluid on the ultrasound scan mimicking the view of a snow-storm in the third-trimester pregnant women is a cause of concern in antenatal management. that high-density intra-amniotic particles were possibly related to vernix caseosa, intra-amniotic bleeding, and meconium.

Although the most commonly reported cause of particulate or echogenic amniotic fluid was vernix caseosa, the reason for concern for the obstetricians in the case of intra-amniotic particles is its potential relationship with meconium as well as fetal compromise

. Free-floating dense particles in the amniotic fluid were also related to lung maturity and it was hypothesized that the source of these particles could be different in each trimester. The concerns for the presence of meconium-stained amniotic fluid in the case of an amniotic sludge may lead the obstetricians to elective induction in term pregnancies before the labor starts spontaneously which also increases the potential complications and caesarean rate

ELIGIBILITY:
Inclusion Criteria:

1. Pregnant women aged between 20, 35 years.
2. Near or Full-term pregnant women admitted for delivery.
3. Reliable date of LMP.
4. Delivered vaginally after spontaneous onset of labor or CS.

Exclusion Criteria:

1. Fetal congenital anomaly by ultrasound (anencephaly& Down syndrome), IUGR or macrosomic fetuses.
2. Multifetal pregnancy.
3. Maternal co-morbidity (Diabetes mellitus, hypertension, cardiac diseases, renal diseases & hemorrhagic diseases) .
4. Maternal infection (Toxoplasmosis, Varicella zoster infection,…).
5. Placental abnormality (abruption placenta & placenta previa)
6. Cases with normal amniotic fluid study with ultrasonography.

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 200 (Actual)
Dates: Start 2022-08-01 (Actual); Primary Completion 2023-08-01 (Actual); Study Completion 2023-08-30 (Actual)

PRIMARY OUTCOMES:
Pregnant females with Echogenic Amniotic Fluid . | At the time of the Delivery
  Estimation the gestational age and neonatal status.

CONTACTS AND LOCATIONS:
Locations (1):
- Al-Azhar University hospitals, Asyut, Egypt